CLINICAL TRIAL: NCT03156166
Title: Distance From the Glottis to the Grille in Children: Ambu AuraGainTM , I-gel, Air-Q Intubating Laryngeal Airway as Intubation Conduits
Brief Title: Distance From the Glottis to the Grille in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: H1704-133-848
Record Dates: First submitted 2017-05-15; First posted 2017-05-17 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: General Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ambu AuraGain (Experimental): Ambu AuraGain is inserted in children undergoing general anesthesia. The size of AuraGain is as follows: size 1 for children <5 kg, size 1.5 for 5-10kg, size 2 for 10-20kg, size 2.5 for 20-30kg. Fiberoptic bronchoscope will be performed to measure the distance between the grill and vocal cord.
  Interventions: Procedure: fiberoptic bronchoscope
- I-gel (Experimental): I-gel is inserted in children undergoing general anesthesia. The size of I-gel is as follows: size 1 for children weighing 2-5kg, size 1.5 for 5-12kg, size 2 for 10-25kg, size 2.5 for 25-35kg. Fiberoptic bronchoscope will be performed to measure the distance between the grill and vocal cord.
  Interventions: Procedure: fiberoptic bronchoscope
- Air-Q intubating laryngeal airway (ILA) (Experimental): Air-Q ILA is inserted in children undergoing general anesthesia. The size of Air-Q ILA is as follows: size 1 for children between 4-7 kg, size 1.5 for 7-17kg, size 2 for 17-30kg, size 2.5 for 30-50kg. Fiberoptic bronchoscope will be performed to measure the distance between the grill and vocal cord.
  Interventions: Procedure: fiberoptic bronchoscope

INTERVENTIONS:
Procedure: fiberoptic bronchoscope — Distance from grille (the end of shaft in supraglottic airway) to glottis is measured using FOB
  Other Names: FOB

SUMMARY:
Ambu AuraGain, I-gel, Air-Q intubating laryngeal airway are the most commonly used supraglottic airway. In children, they can be used as intubation conduits. However, there has been no guideline for optimal insertion depth of endotracheal tube through those supraglottic airway. In this study, the investigators will measure the distance from grille of those supraglottic airways to glottis using fiberoptic bronchoscope in children undergoing anesthesia. This distance allows us to predict an appropriate depth of endotracheal tube when it should be inserted through each supraglottic airway.

ELIGIBILITY:
Inclusion Criteria:

* children < 7 years old undergoing elective surgery

Exclusion Criteria:

* difficult airway
* BMI> 30kg/m2
* emergency operation
* cervical spine disease
* history of esophageal disease and surgery

Max Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 89 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
The distance from grille to glottis | 30 seconds after each supraglottic airway insertion
  The distance from grille to glottis is measured using fiberoptic bronchoscopy

SECONDARY OUTCOMES:
FOB view | 30 seconds after each supraglottic airway insertion
  score 1: no visible glottis, score 2: visible glottis and anterior epiglottis, score 3: visible glottis and posterior epiglottis, and score 4: only glottis visible
Ventilation score | 30 seconds after each supraglottic airway insertion
  no air leak in airway pressure of 15 cmH2O / bilateral chest wall movement/ normal waveform of capnography

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lee JH, Park S, Jang YE, Kim EH, Kim HS, Kim JT. The distance between the glottis and the cuff of a tracheal tube placed through three supraglottic airway devices in children: A randomised controlled trial. Eur J Anaesthesiol. 2019 Oct;36(10):721-727. doi: 10.1097/EJA.0000000000001070. PMID 31415305